CLINICAL TRIAL: NCT00312546
Title: Inhibiting Histone Deacetylase: Toward Eradication of HIV
Brief Title: Study of Valproic Acid to Treat HIV Infected Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: U01AI067854-02 (NIH); CID 0703; 7R01AI064074-01A1 (NIH); 7R01AI045297-08 (NIH); U01A125868
Record Dates: First submitted 2006-04-06; First posted 2006-04-10 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: HIV Infections
Keywords: Virus Latency; Valproic Acid; Histone Deacetylase
MeSH Terms: conditions — HIV Infections | interventions — Enfuvirtide; Valproic Acid

ARMS (4):
- 2A (Experimental): Discontinuation of VPA and enfuvirtide administered for 24 weeks. As of 05/20/08 this step was discontinued.
  Interventions: Drug: Enfuvirtide
- 2B (Experimental): Continuation of VPA for up to 96 weeks. As of 05/20/08 this step was discontinued.
  Interventions: Drug: Valproic acid
- 3A (Experimental): VPA may be added to enfuvirtide for 16 weeks. VPA and enfuvirtide will be continued for up to 96 weeks in responders, and the study will be discontinued in nonresponders.
  Interventions: Drug: Enfuvirtide; Drug: Valproic acid
- 3B (Experimental): Enfuvirtide may be continued for up to 96 weeks. As of 05/20/08 this step was discontinued.
  Interventions: Drug: Enfuvirtide

INTERVENTIONS:
Drug: Enfuvirtide — 90 mg subcutaneously twice daily
  Other Names: T-20
  Arms: 2A; 3A; 3B
Drug: Valproic acid — 500 to 750 mg, taken orally twice daily
  Arms: 2B; 3A

SUMMARY:
A histone deacetylase (HDAC) inhibitor is a class of drug that interferes with the function of HDAC, an enzyme that hides HIV within inactive CD4 cells. These drugs are normally used to treat seizures and other nervous system problems but have been found to work against HIV. The purpose of this study is to investigate the efficacy of valproic acid (VPA), an HDAC inhibitor, in treating HIV infected adults using anti-HIV drugs.

DETAILED DESCRIPTION:
VPA is a type of medication normally used to treat seizures and other nervous system problems. It has been found that VPA works against HIV by releasing the virus from resting CD4 cells, allowing other anti-HIV medications to attack it. The purpose of this study is to assess the efficacy of VPA when used in HIV infected participants using highly active antiretroviral therapy (HAART). The expected duration of participation for individually enrolled participants will depend on which study group the participant is placed in but may range from approximately 24 to 144 weeks.

An initial screening visit will occur about 30 to 120 days prior to study entry. A physical exam, medical and medication history assessment, and blood and urine collection will occur at screening. Leukapheresis and genital secretion collection will occur once 30 to 120 days prior to study entry, separate from the initial screening.

In Step 1, all participants will receive VPA while continuing their current HAART. Doses of VPA will vary by participant. Study visits will occur on Days 0 and 3 and Weeks 1, 2, 4, 8, 12, 16, and 24. A physical exam and blood and urine collection will occur at most visits. Leukapheresis and genital secretion collection will occur at study entry and Weeks 12 and 16. After 24 weeks, participants will enter Step 2. Those participants not responding to VPA in Step 1 will enroll in Step 2A. Participants responding to VPA in Step 1 will enroll in Step 2B.

In Step 2A, participants will discontinue VPA and will receive intensified therapy (enfuvirtide) administered for 24 weeks twice daily. Study visits will occur at Weeks 25, 28, 32, 36, 40, and 48. A physical exam and blood and urine collection will occur at all visits. Leukapheresis will occur at Weeks 36 and 40. Participants who do not respond to intensified therapy in Step 2A will enroll in Step 3A. Participants who respond to intensified therapy in Step 2A will enroll in Step 3B.

In Step 2B, participants will continue to receive VPA for up to 96 weeks. Study visits will occur every 8 weeks until Week 120. A physical exam and blood and urine collection will occur at each visit. Leukapheresis will occur once between Week 72 and Week 120.

In Step 3A, VPA will be added to enfuvirtide for 16 weeks. The study will be discontinued for participants who do not respond. Study visits will occur at screening, entry, Day 0, and Weeks 1, 2, 4, 8, 12, 16, and 22. A physical exam and blood and urine collection will occur at all visits. Leukapheresis will occur after screening, at entry, Day 0 and Weeks 12 and 16.

In Step 3B, participants may continue receiving enfuvirtide for up to 96 weeks. Study visits will occur every 8 weeks until Week 144. A physical exam and blood and urine collection will occur at each visit. Leukapheresis will occur at Week 96 or 144.

Participants may choose to enter an observational period at any time before they start Step 2 or Step 3. During the observational period, participants continue to take HAART but not VPA or enfuvirtide. Upon entering an observational period, study staff will contact the participant every 8 weeks for a review of their medical records. Each participant will have a study visit within 8 weeks of beginning a new step. These interim study screenings include a physical exam, medical history, and blood and urine collection. Participants may be asked to have additional leukapheresis performed if they have discontinued study medications for 12 weeks or more.

Each leukapheresis procedure will take place at the University of North Carolina Apheresis Clinic in Chapel Hill, North Carolina. This study will not provide participants' current HAART regimen medications.

NOTE: As of 05/20/08, the observational period and Steps 1, 2, 2A, 2B, and 3B were discontinued.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected
* Adherent to current HAART regimen
* Adequate vascular access for leukapheresis
* Receiving HAART, defined as at least two nucleoside reverse transcriptase inhibitors plus at least one protease inhibitor or non-nucleoside reverse transcriptase inhibitor, without changes to the regimen within 24 weeks of study entry
* Viral load more than 50 copies/ml on two consecutive occasions for more than 6 months, and less than 200 copies/ml on occasion for more than 6 months prior to study entry
* CD4 count more than 300 cells/mm3
* Willing and able to comply with all study requirements
* Willing to use acceptable forms of contraception

Exclusion Criteria:

* Currently receiving zidovudine or enfuvirtide
* Require certain medications known to interact with valproate (e.g., lamotrigine; barbiturates; carbamazepine; prescription dosages of salicylates, hydantoins, felbamate, and clonazepam)
* Any medical, psychiatric, or job-related responsibility that would interfere with the study. More information about this criterion can be found in the protocol.
* Contraindications to taking VPA (e.g., pregnancy, bleeding disorders, history of pancreatitis, history of hepatitis)
* Receiving interferon, other immunomodulators, or other experimental medications
* Abnormal liver enzyme tests
* Hepatitis B virus infected
* Symptoms of hepatic decompensation
* Blood transfusions or hematopoietic growth factors within 90 days prior to study entry
* Systemic cytotoxic chemotherapy, investigational agents, or immunomodulators within 90 days prior to study entry
* Current drug or alcohol abuse that, in the opinion of the site investigator, would interfere with the study
* Serious illness requiring systemic treatment or hospitalization within 90 days prior to study entry
* Treatment for a current AIDS-defining opportunistic infection within 90 days prior to screening
* Anemic
* Involuntarily incarcerated for treatment of either a psychiatric illness or physical illness (e.g., infectious disease)
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-06; Primary Completion 2009-04 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Frequencies of replication-competent HIV detected in resting CD4 cells | At pre-entry and Week 0 to Weeks 12 and 16

SECONDARY OUTCOMES:
Change in integrated proviral genomes | Throughout study
Genital tract proviral DNA and viral load | Throughout study
Detectable viral load during VPA therapy and if it remains undetectable after VPA is discontinued | Throughout study
HIV-specific antibody changes and CTL responses | From Week 0 to 16
Change in replication-competent HIV detected in resting CD4 cells in study participants after intensified HAART, and after extended VPA therapy with or without intensified HAART | Throughout study
Changes in viral load after intensification of HAART with or without VPA | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: David M. Margolis, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Memorial Hospital, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Jiang G, Espeseth A, Hazuda DJ, Margolis DM. c-Myc and Sp1 contribute to proviral latency by recruiting histone deacetylase 1 to the human immunodeficiency virus type 1 promoter. J Virol. 2007 Oct;81(20):10914-23. doi: 10.1128/JVI.01208-07. Epub 2007 Aug 1. PMID 17670825
- [Background] Siliciano JD, Lai J, Callender M, Pitt E, Zhang H, Margolick JB, Gallant JE, Cofrancesco J Jr, Moore RD, Gange SJ, Siliciano RF. Stability of the latent reservoir for HIV-1 in patients receiving valproic acid. J Infect Dis. 2007 Mar 15;195(6):833-6. doi: 10.1086/511823. Epub 2007 Jan 30. PMID 17299713
- [Background] Smith SM. Valproic acid and HIV-1 latency: beyond the sound bite. Retrovirology. 2005 Sep 19;2:56. doi: 10.1186/1742-4690-2-56. PMID 16168066